CLINICAL TRIAL: NCT05887271
Title: A Multi-Ethnic, Multi-centre raNdomised, Controlled Trial of a Low-energy Diet for Improving Functional Status in Heart Failure With PRESERVED Ejection Fraction (AMEND-preserved)
Brief Title: A Randomised, Controlled Trial of a Low-energy Diet for Improving Functional Status in Heart Failure With PRESERVED Ejection Fraction Preserved Ejection Fraction
Acronym: AMEND
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University of Oxford (Other); University of Manchester (Other); University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0861
Record Dates: First submitted 2023-05-02; First posted 2023-06-02 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Heart Failure, Diastolic; Diabetes Mellitus, Type 2; Diabetes Mellitus Type 2 in Obese; Obesity Adult Onset
Keywords: Heart failure with preserved ejection fraction; Diastolic heart failure; Type 2 diabetes mellitus; Obesity; Meal replacement plan; Cardiac magnetic resonance imaging; Exercise intolerance; Diabetes remission
MeSH Terms: conditions — Heart Failure, Diastolic; Diabetes Mellitus, Type 2; Obesity | interventions — Diet; Diagnostic Imaging; Positron-Emission Tomography; Echocardiography; Hematologic Tests; Electrocardiography; Walk Test

STUDY DESIGN:
Intervention Model Description: Multi-centre, prospective, open-label blinded end-point randomized wait-list controlled trial of low-energy Meal Replacement Plan (MRP) versus guideline-driven care with attention control, and a nested qualitative sub-study.
Masking Description: Participants and investigator will not be blinded to treatment allocation (open label) however, the team analysing the outcomes will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low calorie meal replacement plan (MRP) arm (Experimental): The MRP comprises of 3-4 meals a day (850kcal/day) supplied by Counterweight. Participants will be supported by professional research dieticians, and a study clinician. Participant health and medications will be monitored throughout the study.
  Offered to the comparator arm after 12 weeks as a control participant.
  Interventions: Drug: Low calorie meal replacement plan; Diagnostic Test: Cardiovascular magnetic resonance (CMR) imaging and magnetic resonance spectroscopy; Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Blood test; Diagnostic Test: Electrocardiogram; Diagnostic Test: Accelerometery; Diagnostic Test: 6 minute walk test (6MWT); Diagnostic Test: Skeletal muscle strength using handgrip strength and quadriceps (Cybex dynamometer); Other: Assessment of quality of life and heart failure symptoms; Other: Assessment of sarcopenia; Other: Assessment of frailty; Other: Qualitative interview
- Wait list control arm: Guideline driven care with attention control arm followed by optional MRP (Active Comparator): Dietary advice to participants will be given in line with NICE guidelines for cardiovascular risk modification. Heart failure specific advice on exercise will be given in line with guidelines. After 12 weeks as a control participant, these individuals will then have the option to receive the meal replacement plan and repeat assessments after a further 12 weeks.
  Interventions: Drug: Low calorie meal replacement plan; Diagnostic Test: Cardiovascular magnetic resonance (CMR) imaging and magnetic resonance spectroscopy; Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Blood test; Diagnostic Test: Electrocardiogram; Diagnostic Test: Accelerometery; Diagnostic Test: 6 minute walk test (6MWT); Diagnostic Test: Skeletal muscle strength using handgrip strength and quadriceps (Cybex dynamometer); Other: Assessment of quality of life and heart failure symptoms; Other: Assessment of sarcopenia; Other: Assessment of frailty; Other: Qualitative interview

INTERVENTIONS:
Drug: Low calorie meal replacement plan — Meal replacement diet containing ~850 kcal/day (40% protein, 50% carbohydrate, 10% fat) supplied by Counterweight® (www.counterweight.org).The meal replacement plan will comprise of 3-4 meal packs/day (to equate to 850 kcal) with sweet and savoury options, and an allowance of 100ml semi-skimmed milk or a non-dairy alternative.
  Other Names: Diet
Diagnostic Test: Cardiovascular magnetic resonance (CMR) imaging and magnetic resonance spectroscopy — CMR scanning performed on a 3T MRI scanner. Standardised protocol incorporating cine functional assessment to determine LV mass, systolic function and left atrial volumes; global systolic strain and diastolic strain rates will be assessed by tagging and with tissue tracking analysis from cine images, adenosine rest and stress myocardial perfusion to assess reserve index and qualitative perfusion defects as previously described, aortic distensibility and pulse wave velocity to measure aortic stiffness, delayed contrast enhancement for assessment of LV fibrosis and evidence of previous myocardial infarction. Myocardial and liver triglyceride content will be assessed using the modified Hepafat® sequence or 1H MR spectroscopy at the inter ventricular septum. DIXON technique for the quantification of visceral adiposity and subcutaneous adipose tissue. Cardiac 31P magnetic resonance spectroscopy imaging to assess cardiac muscle energetics according to a standardised operating procedure
  Other Names: CMR
Diagnostic Test: Transthoracic echocardiography — Comprehensive transthoracic echocardiography, including: tissue Doppler indices of diastolic filling and speckle tracking for systolic and diastolic strain/strain rate, exclusion of valvular abnormalities, assessment of LV size and function
Diagnostic Test: Blood test — Collection of blood samples from each participant to characterise the participant's health status and fibroinflammatory markers.
Diagnostic Test: Electrocardiogram — An ECG will be obtained to assess for baseline rhythm.
  Other Names: ECG
Diagnostic Test: Accelerometery — Accelerometer (GeneActiv) measured daily activity levels continuously for 7 consecutive days.
Diagnostic Test: 6 minute walk test (6MWT) — Supervised 6MWT will be performed with symptom assessment using dyspnoea scale (Borg's).
Diagnostic Test: Skeletal muscle strength using handgrip strength and quadriceps (Cybex dynamometer) — Skeletal muscle strength will be measured using a cybex dynamometer.
Other: Assessment of quality of life and heart failure symptoms — Quality of life and HF symptoms will be assessed using the Minnesota Living with Heart Failure (MLWHF) questionnaire, which is used as a standardised measure of self-reported health status, and HF symptoms and is considered to have a good discriminatory power and validity
Other: Assessment of sarcopenia — Participants will be assessed for presence of sarcopenia using the Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls (SARC-F) questionnaire. It is a robust tool for diagnosis of sarcopenia and prediction poor physical function, with excellent specificity in multimorbid individuals.
Other: Assessment of frailty — Frailty will be assessed using the Edmonton Frail Scale (EFS). The EFS is a multidimensional frailty assessment which assesses multiple domains of frailty including functional independence, social support, cognition, medication use, and mood.
Other: Qualitative interview — Participants in the MRP and control groups will be invited to attend a focused semi-structured, 1-2-1 interview aimed to elicit barriers and enablers to the MRP and describe their perspective on the relationship between healthy eating and health interview during the 12-week visit. Participants who complete or drop out will be eligible. Inclusion of participants in the control arm will allow us to compare the experiences of MRP versus health coaching and detect any specific issues people face when trying to introduce lifestyle changes themselves.

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a common and serious complication of obesity and type 2 diabetes (T2D). HFpEF occurs when the heart muscle unable to relax efficiently to pump the blood around the body. This leads to fluid build-up, breathlessness and inability to tolerate physical exertion. People who develop HFpEF do less well because treatment options are limited. Pilot data in patients with obesity and diabetes and a small number of patients with HFpEF have shown improvements in exercise capacity and reversal of changes in the heart and blood vessels. This study will assess if this is achievable in a multi-ethnic cohort of patients with established HFpEF. A total of 63 adults will be invited and allocate by chance into two groups: 1) 12-weeks of a low calorie diet or 2) Standard care and health advice on how to lose weight followed by the option to have the low calorie diet after 12-weeks. The study will determine if weight loss over 12 weeks can improve heart function, symptoms and ability to exercise. Additionally, participants' views on changing their diet and how this has impacted their symptoms will be sought during the study in an optional interview. This will help guide treatments planning in the future to get maximum benefits, and to individualize support to patients from different cultural backgrounds.

DETAILED DESCRIPTION:
Heart failure (HF) with preserved ejection fraction (HFpEF) is a heterogenous syndrome, typified by severe exercise intolerance and with limited treatment options. Weight loss achieved through a low energy meal-replacement plan (MRP) has been shown to lead to reversal of cardiovascular remodelling in ethnically diverse asymptomatic adults with pre-HFpEF and HFpEF. This trial will translate this experience with the pragmatic low energy MRP into a symptomatic, multi-ethnic cohort of obese HFpEF, across four sites (Leicester, Manchester, Leeds and Oxford) to assess its efficacy in improving exercise intolerance, symptoms, quality of life, cardiovascular remodelling, and skeletal myopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Established clinical diagnosis of heart failure with preserved ejection fraction HFpEF (EF>45%) made by a cardiologist or a primary care physician with heart failure expertise, or a heart failure nurse
2. Clinically stable for ≥ 3 months (no admissions to hospital)
3. Obesity (BMI ≥30kg/m2 if white European or ≥27kg/m2 if Asian, Middle Eastern or Black ethnicity)
4. Age ≥18

Exclusion Criteria:

1. Inability to walk/undertake 6-minute walk test
2. Inability to follow a low-energy MRP
3. HFpEF due to infiltrative cardiomyopathy (cardiac amyloidosis or sarcoidosis), genetic hypertrophic cardiomyopathy, restrictive cardiomyopathy/pericardial disease or congenital heart disease.
4. Recovered EF (previous EF < 40%) unless reduced EF was in context of tachycardia induced cardiomyopathy (eg AF/Aflutter).
5. Known heritable, idiopathic or drug-induced pulmonary arterial hypertension
6. Severe chronic obstructive pulmonary disease (FEV1< 1.0L)
7. Severe primary valvular heart disease
8. Anaemia (Hb<100g/L)
9. Severe renal disease (eGFR < 30 ml/min/1.73 m2)
10. Weight loss > 5kg in preceding 3 months.
11. Symptomatic gallstones (including biliary colic) or cholecystitis within last 3 months
12. Active substance abuse (drugs or alcohol)
13. History of bariatric surgery in the last 3 years
14. Active illness likely to cause change in weight
15. Women who are pregnant or are considering pregnancy
16. People currently participating in another clinical research trial that is likely to affect diet or weight change.
17. History of a severe mental illness including an eating disorder

17. Individuals with a diagnosis of Type 1 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in the distance walked during 6 minute walk test (6MWT) | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  The primary outcome measure is a change in the distance walked on 6MWT measured in meters

SECONDARY OUTCOMES:
Beneficial reverse cardiovascular remodelling | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  CMR-derived measures of cardiovascular remodelling defined as left ventricular mass/volume ratio
Change in physical activity levels | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  Improvement in physical activity will be determined by change in daily activity as determined accelerometery
Change in upper limb muscle power | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  Change in muscle power will be determined by handgrip strength using fysiometer
Improvement in exercise tolerance | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  This will be assessed by a)change in Borg dyspnoea scale during 6MWT
Improvement in symptoms of heart failure | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  This will be assessed by a change in the Minessota Living with Heart failure score
Change in frailty | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  This will be assessed by a change in the Edmonton frailty questionnaire score
Change in sarcopenia | Assessed at baseline and 12 weeks, optional repeat at 24 weeks
  This will be assessed by a change in the SARC-F questionnaire score
Exploratory outcome: Improving skeletal and cardiac energetics | Baseline and 12 weeks
  31P magnetic resonance spectroscopy: Cardiac PCr/ATP
Exploratory outcome: change in fibroinflammatory biomarker panel | This will be evaluated at baseline and at 12 weeks
  Exploratory analysis of the O-link fibroinflammatory biomarker panel to identify potential pathways involved in the development, progression or outcomes of HFpEF.

CONTACTS AND LOCATIONS:
Overall Officials: Gerry P McCann, MD, Principal Investigator — University of Leicester
Locations (3):
- United Kingdom (3):
  - University of Leicester, Glenfield Hospital, Groby Road, Leicester, Leicestershire
  - University of Manchester, Wythenshawe Hospital, Southmoor Road, Manchester
  - University of Oxford, John Radcliffe Hospital, Headley Way, Oxford

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Derived] Bilak JM, Squire I, Wormleighton JV, Brown RL, Hadjiconstantinou M, Robertson N, Davies MJ, Yates T, Asad M, Levelt E, Pan J, Rider O, Soltani F, Miller C, Gulsin GS, Brady EM, McCann GP. The Protocol for the Multi-Ethnic, multi-centre raNdomised controlled trial of a low-energy Diet for improving functional status in heart failure with Preserved ejection fraction (AMEND Preserved). BMJ Open. 2025 Jan 28;15(1):e094722. doi: 10.1136/bmjopen-2024-094722. PMID 39880434